CLINICAL TRIAL: NCT06878417
Title: The Effectiveness of Oral Cannabis Extracts for Osteoarthritic Pain: an Internal Pilot, Placebo Controlled, Blinded Randomized Trial
Brief Title: Cannabinoids for Osteoarthritis Pain Effectiveness Trial
Acronym: COPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 24-5572
Record Dates: First submitted 2025-02-24; First posted 2025-03-17 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-05

CONDITIONS: Osteoarthritis of Knee; Osteoarthritis Hip
Keywords: Medical Cannabis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patients, study staff (except the unblinded research assistant who will be preparing and dispensing the IPs), care providers, adjudicators, data analysts, and investigators will be blinded to the active ingredient in the IPs and group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBD (Cannabidiol) (Experimental): Each capsule contains a concentration of 50 mg of Cannabidiol (CBD). Participants will receive CBD for a total duration of 8 weeks.
  Interventions: Drug: CBD
- THC (∆9-tetrahydrocannabinol) (Experimental): Each capsule contains a concentration of 3 mg of ∆9-tetrahydrocannabinol (THC). Participants will receive THC capsules for a total duration of 8 weeks.
  Interventions: Drug: THC
- Placebo (Placebo Comparator): Participants will receive matching placebo capsules for a total duration of 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CBD — The starting dose will be 1 capsule per day (50 mg CBD) taken orally. The dose will be gradually increased over the first four weeks, based on patient assessment, up to a maximum of five capsules per day (250 mg CBD) in divided doses. Once the dose that maximizes potential therapeutic effects while minimizing adverse effects has been determined, it will be maintained for the remaining four weeks of the trial.
  Other Names: AVCN319301a
  Arms: CBD (Cannabidiol)
Drug: THC — The starting dose will be 1 capsule per day (3 mg THC) taken orally. The dose will be gradually increased over the first four weeks, based on patient assessment, up to a maximum of five capsules per day (15 mg THC) in divided doses. Once the dose that maximizes potential therapeutic effects while minimizing adverse effects has been determined, it will be maintained for the remaining four weeks of the trial.
  Other Names: AVCN319301b
  Arms: THC (∆9-tetrahydrocannabinol)
Drug: Placebo — The starting dose will be 1 capsule per day taken orally. The dose will be gradually increased over the first four weeks, based on patient assessment, up to a maximum of five capsules per day in divided doses. Once the dose that maximizes potential therapeutic effects while minimizing adverse effects has been determined, it will be maintained for the remaining four weeks of the trial.
  Arms: Placebo

SUMMARY:
This study aims to investigate whether oral cannabis extracts can effectively manage pain caused by osteoarthritis (OA), a common joint condition affecting one in seven Canadians. Current OA treatments often have limited effectiveness and may cause side effects. As a result, many individuals with OA turn to medical cannabis for pain relief, despite limited scientific evidence supporting its efficacy.

The goal of this study is to assess the feasibility of a larger trial evaluating the effects of two cannabis compounds-CBD and THC-compared to a placebo (a look-alike substance containing no active drug) on pain interference in patients with hip and/or knee osteoarthritis.

Participants will:

* Take either CBD, THC, or a placebo capsule daily for 8 weeks
* Complete follow-ups remotely, with no in-person clinic visits required
* Maintain a diary tracking their study drug usage and any additional pain medications

DETAILED DESCRIPTION:
The rationale for this study lies in the significant impact of osteoarthritis (OA) on individuals and society, coupled with the limited effectiveness and potential side effects of current treatments. OA is a prevalent joint disease affecting one in seven Canadians, causing pain, stiffness, and swelling that can significantly disrupt daily life. The economic burden of OA is substantial, costing Canada an estimated $27.5 billion annually. With no cure for OA, current treatments focus on managing pain, the most disabling symptom, and improving physical function. The study addresses a critical gap in knowledge concerning the use of medical cannabis (MC) for OA pain management. Despite a considerable number of Canadians turning to MC for symptom relief, there is a lack of high-quality evidence supporting its effectiveness. This discrepancy between widespread use and insufficient scientific data creates a pressing need for rigorous research. Surveys indicate that approximately 20% of patients with musculoskeletal pain, including OA, have used or are using MC for pain management. Anecdotal evidence suggests effectiveness for some patients, but the lack of robust data leaves important questions unanswered. Key issues include identifying the optimal type of product, the right dose, and the best mode of administration to maximize effectiveness while minimizing side effects. The study is further motivated by the fact that OA patients often face challenges in obtaining clear guidance from healthcare providers regarding MC use due to the scarcity of evidence and concerns about safety. This lack of guidance may result in misinformation, unnecessary expenses, and potential risks for patients. The rationale is strengthened by strong pre-clinical evidence suggesting that cannabinoids, the active compounds in MC, may effectively address OA pain. These compounds act on cannabinoid receptors and other receptors involved in pain and inflammation pathways within the joints. Given the increasing use of MC for OA pain, the lack of high-quality clinical evidence, and the promising pre-clinical data, the study proposes an internal pilot trial to assess the feasibility of a larger, definitive randomized controlled trial (RCT). The internal pilot aims to optimize recruitment and retention strategies before launching a comprehensive investigation into the effectiveness of specific cannabis compounds (CBD and THC) in managing OA pain.

This pilot study is a multicentre, blinded, randomized, placebo-controlled, 3-arm, parallel group (1:1:1 CBD, THC, placebo) internal pilot trial in patients with hip and/or knee osteoarthritis pain. Patients will receive CBD (intervention), THC (intervention), or placebo (control) for 8 weeks.

The primary objective of this internal pilot RCT is to determine the feasibility of a blinded, randomized, placebo-controlled, 3-arm, parallel group trial of oral cannabinoids for improving pain interference in patients with hip and/or knee osteoarthritis. Specifically, this study will determine whether the planned definitive RCT is feasible with respect to patient enrollment, protocol adherence, and data completeness.

This is a decentralized trial whereby participants will be recruited and enrolled from three sites, but all other study-related activities (e.g., shipping of study product, follow-up assessments, etc.) will be conducted by the central coordinating centre (Anesthesia Clinical Trials Unit (ACTU), a clinical research organization located at Toronto General Hospital (TGH)) remotely without requiring patients to attend in-person study visits.

A total of 100 patients will be recruited across all the sites.

Patients from all the recruiting sites will be followed up at the end of weeks 1, 2, 3, 4, 6, and 8 after treatment initiation by the central coordinating centre (ACTU).

During each follow up assessment:

1. Patients will be assessed for a follow up check-in which includes a brief discussion of treatment efficacy and adverse effects and it will last approximately 10-15 minutes or as long as is needed to address any and all patient concerns. During baseline assessment, the patient receives instructions on starting dose. At 1, 2-, 3- and 4-weeks, the patients will also receive instructions regarding dose titration, as needed.
2. Patients complete the set of questionnaires which which will be sent to them a day prior of their scheduled follow up. The questionnaires will assess pain severity and interference, physical functioning, sleep quality, anxiety, and depression. In addition, all participants will complete a health-related quality of life questionnaire and rate the overall improvement related to the intervention. The questionnaires will be administered via standardized case report forms in a secure online portal (REDCap).
3. The patient will also be followed by the blinded research assistant to complete other study related activities (i.e. assessment of study drug compliance, reiterate the importance of a study drug diary and how data should be recorded, confirms capsules count, study drug diary review etc.)

Patients will be unblinded following their 8-week follow-up, which takes place eight weeks after the initiation of treatment. Those choosing to discontinue the investigational products (CBD and THC) will receive support to taper off and will have scheduled follow-ups at the end of the 10th and 12th weeks to monitor the progress of participants during the tapering phase, and for those who choose to continue using cannabis, assistance will be provided to help them secure their own supply of medical cannabis during the next 4-week period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-80 years
2. Diagnosed with hip and/or knee osteoarthritis as per the American College of Rheumatology criteria
3. Experiencing moderate to severe pain interference as indicated by a PROMIS-PI SF-6a T-score ≥ 60
4. Have not initiated any new analgesics or osteoarthritis treatments in the previous 4 weeks
5. Able to self-report, understand and read English or French

Exclusion Criteria:

1. Hip or knee surgery planned in the coming 4 months,
2. Injection into the affected joint(s) within the past 3 months (e.g., cortisone, plasma-rich protein, etc.),
3. Planned injection into the affected joint(s) during trial period,
4. Inflammatory arthritis (e.g., rheumatoid arthritis, Psoriatic arthritis, gout, etc.),
5. Contraindications to taking cannabis/cannabinoids,
6. Used nabilone or nabiximols in the last 30 days,
7. Used cannabis (medical or recreational) in the last 30 days (to allow sufficient washout),
8. A history of diagnosed cannabis use disorder or dependence,
9. Active substance use disorder,
10. Current DSM-V diagnosis of bipolar disorder, major depression, or psychosis,
11. An uncontrolled medical or major psychiatric disorder,
12. Currently on warfarin,
13. Known pregnancy or currently breastfeeding,
14. Men and women planning a pregnancy during the study or in the 12 weeks after stopping IPs
15. No fixed address or a plan to change addresses in the coming 4 months,
16. Known or suspected allergy to palm/coconut oil

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility outcome: pertaining to the enrollment rate | Through study completion, an average of 1 year
  Percentage of eligible and interested patients enrolled
Feasibility outcome: pertaining to the Protocol adherence | Up to 8 weeks post-treatment
  Percentage of participants with no major protocol deviation (i.e., no concomitant cannabis use or initiation of new OA treatment)
Feasibility outcome: pertaining to data completeness | Up to 8 weeks post-treatment
  Percentage of enrolled participants with complete PROMIS Pain Interference data at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Hance Clarke, MD, Principal Investigator — University Health Network, Toronto
Locations (3):
- Canada (3):
  - University Health Network, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - McGill University Health Centre/Montreal General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No